CLINICAL TRIAL: NCT05567887
Title: A PHASE I, OPEN LABEL STUDY TO EVALUATE THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF TTI-622 (PF-07901801), A SINGLE AGENT IN JAPANESE PARTICIPANTS WITH RELAPSED OR REFRACTORY LYMPHOMA
Brief Title: A Study to Learn About the Study Medicine (Called Maplirpacept (PF-07901801)) in Japanese With Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4971009
Record Dates: First submitted 2022-09-22; First posted 2022-10-05 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Lymphoma; Multiple Myeloma
Keywords: Lymphoma; multiple myeloma; maplirpacept; TTI-622; PF-07901801; C4971009; Phase 1; Japan
MeSH Terms: conditions — Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- maplirpacept (PF-07901801) (Experimental): maplirpacept (PF-07901801)
  Interventions: Drug: maplirpacept (PF-07901801)

INTERVENTIONS:
Drug: maplirpacept (PF-07901801) — maplirpacept (PF-07901801)
  Other Names: TTI-622

SUMMARY:
The purpose of this clinical trial is to learn about how safe and tolerable is the study medicine (called maplirpacept (PF-07901801)) when taken for the treatment of lymphoma or multiple myeloma (a type of cancer that affects your body's infection-fighting cells, lymphocytes or plasma cell).

This study is seeking participants who:

* are 18 years of age or older
* have worsening and difficult to manage type of lymphoma or multiple myeloma
* Have adequately functioning organs
* are not on long term use of steroids which are given either by mouth or as shots
* have no major heart related disease etc.

All participants in this study will receive maplirpacept (PF-07901801) as an IV infusion (given directly into a vein) at the study clinic every week.

Participants will continue to receive maplirpacept (PF-07901801) until their progress of cancer worsens or the participants do not wish to take the study medicine.

The experiences of the people receiving the study medicine will be collected. This will help to understand if the study medicine maplirpacept (PF-07901801), is safe and can be given to Japanese people.

DETAILED DESCRIPTION:
CD47 is a cell-surface protein expressed on multiple normal cell types and often at high levels on many malignant tumor cells. Maplirpacept (PF-07901801) is a soluble recombinant fusion protein created by directly linking the sequences encoding the CD47 binding domain of human Signal Regulatory Protein alpha with the fragment crystallizable domain of human Immunoglobulin 4. maplirpacept (PF-07901801) functions as a soluble decoy receptor, preventing CD47 from delivering its antiphagocytic signal. Neutralization of the inhibitory CD47 signal enables macrophage activation and anti-tumor effects by pro-phagocytic signals present on the tumor cells.

The objective of this study is to confirm safety and tolerability of single agent maplirpacept (PF-07901801) at the recommended phase 3 dose in Japanese participants with relapsed or refractory lymphoma or multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory lymphoma (Hodgkin's or non-Hodgkin's) or multiple myeloma
* Disease must have progressed with standard anticancer therapies
* measurable disease
* Capable of giving signed informed consent
* Eastern cooperative oncology group performance status 0 or 1
* Adequate organ functions

Exclusion Criteria:

* Known, current central nervous system or interstitial lung disease involvement
* History of hemolytic anemia or positive direct antiglobulin test or active bleeding disorder
* Chronic use of systemic corticosteroids of more than 20 mg/day of prednisone or equivalent
* Significant cardiovascular disease
* Other significant medical condition unrelated to the primary malignancy
* Radiation therapy within 14 days of study treatment administration
* Hematopoietic stem cell transplant within 90 days before the planned start of study treatment
* Antiplatelet/anticoagulant agents within 14 days before planned start of study treatment
* Patients sustaining major surgery at least 4 weeks prior to study enrollment
* Use of any investigational agent or any anticancer drug within 14 days before planned start of study treatment
* Prior anti-CD47 and anti-Signal Regulatory Protein alpha therapy
* Active, uncontrolled bacterial, fungal, or viral infection
* Investigator site staff directly involved in the conduct of the study and their family members

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity (DLT) in lymphoma | up to 21 days
  Number of participants with DLTs

SECONDARY OUTCOMES:
Number of adverse events as characterized by type | Through study completion, up to 18 months
  overall safety profile of maplirpacept (PF-07901801)
Number of adverse events as characterized by frequency | Through study completion, up to 18 months
  overall safety profile of maplirpacept (PF-07901801)
Number of adverse events as characterized by severity | Through study completion, up to 18 months
  overall safety profile of maplirpacept (PF-07901801)
Number of adverse events as characterized by timing | Through study completion, up to 18 months
  overall safety profile of maplirpacept (PF-07901801)
Number of adverse events as characterized by relationship to maplirpacept (PF-07901801) | Through study completion, up to 18 months
  overall safety profile of maplirpacept (PF-07901801)
Number of adverse events as characterized by seriousness | Through study completion, up to 18 months
  overall safety profile of maplirpacept (PF-07901801)
Number of participants with clinically significant change from baseline in laboratory abnormalities as characterized by type | Through study completion, up to 18 months
  overall safety profile of maplirpacept (PF-07901801)
Number of participants with clinically significant change from baseline in laboratory abnormalities as characterized by frequency | Through study completion, up to 18 months
  overall safety profile of maplirpacept (PF-07901801)
Number of participants with clinically significant change from baseline in laboratory abnormalities as characterized by severity | Through study completion, up to 18 months
  overall safety profile of maplirpacept (PF-07901801)
Number of participants with clinically significant change from baseline in laboratory abnormalities as characterized by timing | Through study completion, up to 18 months
  overall safety profile of maplirpacept (PF-07901801)
Number of participants with severe thrombocytopenia and anemia in R/R multiple myeloma | Through study completion, up to 18 monghs
  overll safety profile of maplirpacept (PF-07901801)
maximum observed concentration, steady state (ss) of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
time to maximum concentration,ss of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
area under the curve last,ss of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
area under the curve tau,ss of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
time to maximum concentration of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
trough concentration of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
area under the curve last of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
clearance of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
area under the curve tau of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
volume of distribution at steady-state of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
area under the curve tau,ss/area under the curve tau,sd of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
area under the curve inf of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
terminal elimination half-life off maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
maximum observed concentration of maplirpacept (PF-07901801) | Through study completion, up to 18 months
  pharmacokinetics of maplirpacept (PF-07901801)
Incidence and titers of anti-drug antibodies against maplirpacept (PF-07901801) | Through study completion, up to 18 months
  immunogenicity of maplirpacept (PF-07901801)
Incidence and titers of neutralizing antibodies against maplirpacept (PF-07901801) | Through study completion, up to 18 months
  immunogenicity of maplirpacept (PF-07901801)
overall response rate | From date of registration until the date of first documented progression or date of death from any cause, cause, whichever comes first, assessed up to 18 months
  preliminary antitumor activity of maplirpacept (PF-07901801)
progression free survival | From date of registration until the date of first documented progression or date of death from any cause, cause, whichever comes first, assessed up to 18 months
  preliminary antitumor activity of maplirpacept (PF-07901801)
time to response | From date of registration until the date of first documented progression or date of death from any cause, cause, whichever comes first, assessed up to 18 months
  preliminary antitumor activity of maplirpacept (PF-07901801)
duration of response | From date of registration until the date of first documented progression or date of death from any cause, cause, whichever comes first, assessed up to 18 months
  preliminary antitumor activity of maplirpacept (PF-07901801)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Japan (4):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4971009